CLINICAL TRIAL: NCT05927337
Title: Cognitive-Behavioral Therapy for Managing Obesity in People With Chronic Kidney Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Medical Centre Ljubljana (Other)
Collaborators: Slovenian Research Agency (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: L3-KKM-MR
Record Dates: First submitted 2023-05-30; First posted 2023-07-03 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-05

CONDITIONS: Chronic Kidney Diseases; Obesity; Overweight
Keywords: Obesity; Chronic KIdney Disease; Overweight; Cognitive Behavioral Therapy; Weight loss; Weight maintenance
MeSH Terms: conditions — Renal Insufficiency, Chronic; Obesity; Overweight; Weight Loss | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Masking Description: The nature of the intervention (Cognitive Behavioral Therapy) makes it impossible to mask interventions assigned.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Behavioral Therapy for managing Obesity (Experimental): Participants will be enrolled in a 4-month programme of cognitive behavioural therapy for obesity management. The programme is described in more detail in the annex. The programme will consist of 12 individual sessions, with weekly sessions for the first eight weeks and bi-monthly sessions for the following eight weeks.
  Treatment as usual: participants will receive three sessions with a dietician to receive basic information on appropriate diet, energy deficit and nutrition plan and three sessions with a kinesiologist to receive advice on physical activity.
  Interventions: Behavioral: Cognitive Behavioral Therapy (CBT) for managing Obesity
- Control group (No Intervention): Treatment as usual: participants will receive three sessions with a dietician to receive basic information on appropriate diet, energy deficit and nutrition plan and three sessions with a kinesiologist to receive advice on physical activity.

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy (CBT) for managing Obesity — Patients included in the intervention group will be treated with a tailored cognitive behavioural therapy programme for obesity management. The programme is designed and adapted from the Individualised Cognitive Behavioural Therapy for Obesity Management programme (Dalle Grave et al., 2018), which is divided into six content modules aimed at weight loss and weight maintenance. For the purpose of the research, an abbreviated programme will be designed and used, and the content modules will remain the same as in the original version of the programme.
  Arms: Cognitive Behavioral Therapy for managing Obesity

SUMMARY:
In the study Cognitive-Behavioral Therapy (CBT) for Managing Obesity in People with Chronic Kidney Disease (CKD) the investigators will test whether CBT programme is effective for weight loss and weight maintenance after the treatment programme in patients with obesity, chronic kidney disease and proteinuria. The investigators will test whether subjects randomised to the intervention group and receiving cognitive behavioural therapy can achieve greater weight loss and proteinuria reduction in chronic kidney disease than subjects randomised to the control group and not receiving cognitive behavioural therapy. Both groups of subjects will be counselled by a dietician to improve their diet and reduce excess weight and to kinesiologist for advice on physical activity.

DETAILED DESCRIPTION:
The inclusion of clinical psychological and psychotherapeutic interventions in the management of overweight and obese patients can contribute significantly to the success of lifestyle changes and higher motivation for weight loss. Indeed, cognitive processes play an important role in the maintenance of dysfunctional eating patterns. Cognitive-behavioural therapy and behavioural therapies are widely used in the weight loss process. The starting point of behavioural and cognitive-behavioural therapies is that behaviours are learned and therefore can be unlearned, changed or replaced through a therapeutic process involving a variety of behavioural and cognitive techniques.

Individualised cognitive-behavioural therapy for obesity management has three central goals, namely i) losing and maintaining an appropriate weight, ii) adopting and maintaining a lifestyle that allows for appropriate weight control, and iii) developing a stable mindset about weight control. In the therapeutic process, the therapist develops a collaborative relationship with the patient, in which the patient plays an active role in abandoning unhealthy lifestyle habits and developing more appropriate ones that facilitate the achievement and maintenance of a healthy weight. The approach has been designed for different levels of obesity, is delivered in an individual or group format and includes a preparatory phase (one to two sessions) in which the level of obesity, associated medical and psychological problems are assessed and the patient is engaged in the treatment, followed by a first phase, focused on weight loss, and a second phase, focused on weight maintenance.

The content of the programme includes behavioural strategies to help weight loss and environmental modification, cognitive techniques and techniques to prevent weight regain. The treatment programme will consist of 12 sessions spread over four months. The initial sessions will focus on weight loss, while the later sessions will focus on consolidation or learning strategies for weight maintenance.

Obesity is one of the common health problems encountered by patients with chronic kidney disease. By making lifestyle changes and reducing weight, individuals can achieve a slower disease progression and a better quality of life. Knowledge in this area would be useful for the planning of clinical psychological and medical management of patients with chronic kidney disease and would also shed light on the role of the psychologist in the management of this patient population.

The specific objectives of the study are:

* To investigate the effectiveness of an individualised cognitive behavioural therapy programme for the management of obesity in patients with chronic kidney disease.
* To analyse the association of psychological variables with the effectiveness of a cognitive-behavioural intervention.
* Analysis of the impact of a cognitive behavioural intervention for obesity management on quality of life, depression and anxiety.

ELIGIBILITY:
Inclusion Criteria:

* patients with chronic kidney disease (proteinuric form) from stage 2 to stage 4 (oGF 60 to 15 ml/min/1.73m2);
* with or without associated type 2 diabetes mellitus;
* with a body mass index greater than 30 kg/m2 or waist circumference greater than 94 cm (men) or 80 cm (women);
* who have an estimated daily proteinuria exceeding 200 mg protein per g urinary creatinine.

Exclusion Criteria:

* acute psychiatric illness or chronic, poorly managed psychiatric illness;
* dementia;
* bioimpedance findings of low lean body mass index below that expected for age and sex (or presence of any other sarcopenic obesity criteria);
* active chronic inflammatory disease (e.g. active vasculitis, SLE, rheumatoid arthritis) or active cancer;
* active nephrotic syndrome;
* NYHA grade 3 or 4 heart failure;
* spontaneous weight loss of 5% or more in the last 6-month period;
* receiving induction immunosuppression therapy for autoimmune renal disease (receiving maintenance immunosuppression therapy for no retention);
* any other clinical factor that puts the patient at risk with regard to metabolic stability and daily energy expenditure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Body Mass Index (BMI) | baseline, 4 months, 7 months, 12 months
  derived from the mass and height of a person
Change in Proteinuria | baseline, 4 months, 7 months, 12 months
  daily proteinuria exceeding 200 mg protein per g creatinine in urine

SECONDARY OUTCOMES:
Change in Waist circumference | baseline, 4 months, 7 months, 12 months
  in centimeters
Change in Body Fat Percentage | baseline, 4 months, 7 months, 12 months
  measured with bioelectrical impedance analysis
Change in Cholesterol | baseline, 4 months, 7 months, 12 months
  LDL Cholesterol level
Change in Systolic and Diastolic Blood Pressure | baseline, 4 months, 7 months, 12 months
  pressure of circulating blood against the walls of blood vessels
Change in Blood Sugar | baseline, 4 months, 7 months, 12 months
  blood sugar concentration - measure of glucose concentrated in the blood
Chanhe in Glycated Haemoglobin | baseline, 4 months, 7 months, 12 months
  est shows an average of the blood sugar level over the past 90 days and represents a percentage.
Change in Depression | baseline, 4 months, 7 months, 12 months
  Measured with Beck Depression Inventory; scores 0-9: indicates minimal depression 10-18: indicates mild depression 19-29: indicates moderate depression 30-63: indicates severe depression.
Change in Anxiety | baseline, 4 months, 7 months, 12 months
  Measured with The State-Trait Anxiety Inventory. The total score ranges from 0-63. The following guidelines are recommended for the interpretation of scores: 0-9, normal or no anxiety; 10-18, mild to moderate anxiety; 19-29, moderate to severe anxiety; and 30-63, severe anxiety.
Change in Quality of Life measure | baseline, 4 months, 7 months, 12 months
  Measured with SF-36v2®. The SF-36v2® Health Survey measures functional health and well-being from the patient's perspective with questions that span eight health domains: physical functioning, role-physical, bodily pain, general health, vitality, social functioning, role-emotional and mental health. To score the SF-36, scales are standardized with a scoring algorithm or by the SF-36v2 scoring software to obtain a score ranging from 0 to 100. Higher scores indicate better health status, and a mean score of 50 has been articulated as a normative value for all scales.
Risk Factors for Eating Disorders | baseline, 4 months, 7 months, 12 months
  Measured with Eating disorder Examination Questionnaire (EDEQ-6). EDE-Q is a 28-item self-report questionnaire. The EDE-Q is scored using a 7-point, forced-choice rating scale (0-6) with scores of 4 or higher indicative of clinical range. The subscale and global scores reflect the severity of eating disorder psychopathology.
Personality Traits | baseline
  Measured with Big Five Questionnaire BFQ. The BFQ was designed to assess the constellation of traits defined by the Five Factor Theory of Personality. It consist of 132 items using 5-point ratings (1 = very false for me to 5 = very true for me). It has 5 sub-scales (neuroticism, extraversion, openness, agreeableness, and conscientiousness). Higher score means a more pronounced trait.
General Self-Efficacy | baseline
  Measured with General Self-Efficacy Scale GSE. GSE scores range from 10 to 40, where the higher the score, the greater the individual's generalised self-efficacy belief.

CONTACTS AND LOCATIONS:
Overall Officials: Jernej Pajek, PhD, Study Director — Department of Nephrology, University Medical Centre Ljubljana, Ljubljana, Slovenia.; Jadranka Buturovič Ponikvar, PhD, Study Chair — Department of Nephrology, University Medical Centre Ljubljana, Ljubljana, Slovenia.
Locations (1):
- University Medical Centre Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: Yes
It is planned to publish it on the repository of University of Ljubljana. Personal data will not be provided, participants will be encrypted and unrecognizable.
Supporting Information: Study Protocol
Time Frame: After the study will be finished
Access Criteria: Not fully decided yet

REFERENCES:
- [Background] Anderson JW, Konz EC, Frederich RC, Wood CL. Long-term weight-loss maintenance: a meta-analysis of US studies. Am J Clin Nutr. 2001 Nov;74(5):579-84. doi: 10.1093/ajcn/74.5.579. PMID 11684524
- [Background] Comsa L, David O, David D. Outcomes and mechanisms of change in cognitive-behavioral interventions for weight loss: A meta-analysis of randomized clinical trials. Behav Res Ther. 2020 Sep;132:103654. doi: 10.1016/j.brat.2020.103654. Epub 2020 Jun 2. PMID 32683134
- [Background] Conley MM, McFarlane CM, Johnson DW, Kelly JT, Campbell KL, MacLaughlin HL. Interventions for weight loss in people with chronic kidney disease who are overweight or obese. Cochrane Database Syst Rev. 2021 Mar 30;3(3):CD013119. doi: 10.1002/14651858.CD013119.pub2. PMID 33782940
- [Background] Dalle Grave R, Calugi S, Bosco G, Valerio L, Valenti C, El Ghoch M, Zini D. Personalized group cognitive behavioural therapy for obesity: a longitudinal study in a real-world clinical setting. Eat Weight Disord. 2020 Apr;25(2):337-346. doi: 10.1007/s40519-018-0593-z. Epub 2018 Oct 10. PMID 30306498
- [Background] Dalle Grave R, Sartirana M, Calugi S. Personalized cognitive-behavioural therapy for obesity (CBT-OB): theory, strategies and procedures. Biopsychosoc Med. 2020 Mar 9;14:5. doi: 10.1186/s13030-020-00177-9. eCollection 2020. PMID 32175002
- [Background] Dalle Grave R, Sartirana M, El Ghoch M, Calugi S. Personalized multistep cognitive behavioral therapy for obesity. Diabetes Metab Syndr Obes. 2017 Jun 1;10:195-206. doi: 10.2147/DMSO.S139496. eCollection 2017. PMID 28615960
- [Background] Dombrowski SU, Knittle K, Avenell A, Araujo-Soares V, Sniehotta FF. Long term maintenance of weight loss with non-surgical interventions in obese adults: systematic review and meta-analyses of randomised controlled trials. BMJ. 2014 May 14;348:g2646. doi: 10.1136/bmj.g2646. PMID 25134100
- [Background] Greaves CJ, Sheppard KE, Abraham C, Hardeman W, Roden M, Evans PH, Schwarz P; IMAGE Study Group. Systematic review of reviews of intervention components associated with increased effectiveness in dietary and physical activity interventions. BMC Public Health. 2011 Feb 18;11:119. doi: 10.1186/1471-2458-11-119. PMID 21333011
- [Background] Jacob A, Moullec G, Lavoie KL, Laurin C, Cowan T, Tisshaw C, Kazazian C, Raddatz C, Bacon SL. Impact of cognitive-behavioral interventions on weight loss and psychological outcomes: A meta-analysis. Health Psychol. 2018 May;37(5):417-432. doi: 10.1037/hea0000576. PMID 29698017
- [Background] Jansen A, Houben K, Roefs A. A Cognitive Profile of Obesity and Its Translation into New Interventions. Front Psychol. 2015 Nov 27;6:1807. doi: 10.3389/fpsyg.2015.01807. eCollection 2015. PMID 26640451
- [Background] Loveman E, Frampton GK, Shepherd J, Picot J, Cooper K, Bryant J, Welch K, Clegg A. The clinical effectiveness and cost-effectiveness of long-term weight management schemes for adults: a systematic review. Health Technol Assess. 2011 Jan;15(2):1-182. doi: 10.3310/hta15020. PMID 21247515
- [Background] Navaneethan SD, Yehnert H, Moustarah F, Schreiber MJ, Schauer PR, Beddhu S. Weight loss interventions in chronic kidney disease: a systematic review and meta-analysis. Clin J Am Soc Nephrol. 2009 Oct;4(10):1565-74. doi: 10.2215/CJN.02250409. Epub 2009 Sep 17. PMID 19808241
- [Background] Wang Y, Chen X, Song Y, Caballero B, Cheskin LJ. Association between obesity and kidney disease: a systematic review and meta-analysis. Kidney Int. 2008 Jan;73(1):19-33. doi: 10.1038/sj.ki.5002586. Epub 2007 Oct 10. PMID 17928825
- [Derived] Kurnik Mesaric K, Kodric J, Logar Zakrajsek B, Pernat AM, Bogataj S, Pajek J. Cognitive behavioral therapy for managing obesity in patients with chronic kidney disease: Study protocol for a randomized controlled trial. Contemp Clin Trials Commun. 2023 Nov 21;36:101236. doi: 10.1016/j.conctc.2023.101236. eCollection 2023 Dec. PMID 38074489